CLINICAL TRIAL: NCT07364552
Title: Patient-Specific Occlusal Splints Designed Using MODJAW Kinematic Data: A Prospective Clinical Study
Brief Title: Patient-Specific Occlusal Splints Using MODJAW Kinematics
Acronym: MOD-SP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Dr. Merve Benli, Dr, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U-116S697
Record Dates: First submitted 2026-01-12; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Bruxism
Keywords: Occlusal splint
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups: (1) MODJAW-based patient-specific splint group, or (2) standard occlusal splint group. Each participant follows their assigned intervention for 8 weeks. Outcomes are compared between the groups at baseline and post-intervention.
Masking Description: Not applicable; this is an open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MODJAW-Based Patient-Specific Splint (Experimental): Participants receive a patient-specific occlusal splint designed using MODJAW 3D mandibular kinematic data. The splint is fabricated via CAD/CAM and worn according to study instructions for 8 weeks.
  Interventions: Device: MODJAW-Based Patient-Specific Occlusal Splint
- Standard Occlusal Splint (Experimental): Participants receive a conventional occlusal splint fabricated using standard methods. The splint is worn according to study instructions for 8 weeks.
  Interventions: Device: Standard Occlusal Splint

INTERVENTIONS:
Device: MODJAW-Based Patient-Specific Occlusal Splint — A custom occlusal splint designed using MODJAW-recorded 3D mandibular movement data. Fabricated via CAD/CAM to fit the patient's unique jaw movements. Worn nightly (or per instructions) for 8 weeks.
  Arms: MODJAW-Based Patient-Specific Splint
Device: Standard Occlusal Splint — A conventional occlusal splint made using standard methods without patient-specific mandibular movement data. Worn nightly (or per instructions) for 8 weeks.
  Arms: Standard Occlusal Splint

SUMMARY:
This clinical study is designed to evaluate the effectiveness of patient-specific occlusal splints created using MODJAW, a jaw-tracking device that records 3D mandibular movements. Occlusal splints are commonly used to treat bruxism (teeth grinding) and temporomandibular joint (TMJ) disorders, which can cause jaw pain, headaches, and worn teeth. Traditional splints are made using standard designs that do not consider each patient's unique jaw movements.

In this study, 40 participants with mild-to-moderate bruxism or TMJ dysfunction will be randomly assigned to two groups. One group will receive custom splints designed using MODJAW kinematic data, while the other group will receive standard occlusal splints. Participants will use their assigned splint for 8 weeks.

The study will measure:

Jaw movement patterns using MODJAW

TMJ pain levels

Patient comfort and satisfaction

The main goal is to determine whether MODJAW-based, patient-specific splints provide better jaw function, reduced pain, decreased teeth grinding, and higher patient satisfaction compared to standard splints.

Participants will be monitored throughout the study to ensure safety, comfort, and proper splint use. This study is expected to help dentists design more effective, personalized splints in the future and improve treatment outcomes for people with jaw disorders or bruxism.

DETAILED DESCRIPTION:
Detailed Description:

Background and Rationale:

Bruxism and temporomandibular joint (TMJ) disorders are common conditions that can lead to jaw pain, headaches, tooth wear, and impaired quality of life. Occlusal splints are commonly prescribed to manage these conditions by stabilizing the jaw and distributing occlusal forces. Standard splints, however, are typically fabricated using uniform designs that do not account for the individual jaw movement patterns of each patient. Recent advances in digital dentistry, including the use of jaw-tracking devices such as MODJAW, allow clinicians to capture three-dimensional mandibular kinematics in real time. By using this information, occlusal splints can be designed to match the specific movement patterns of each patient, potentially improving comfort, jaw function, and clinical outcomes.

This study aims to evaluate whether patient-specific occlusal splints designed using MODJAW kinematic data provide superior clinical outcomes compared to standard occlusal splints.

Study Objectives:

To compare mandibular movement patterns between MODJAW-based patient-specific splints and standard occlusal splints.

To evaluate the effect of MODJAW-based splints on bruxism frequency and intensity.

To assess TMJ pain reduction in participants using MODJAW-based splints versus standard splints.

To determine patient satisfaction and comfort with patient-specific versus standard splints.

Study Design:

This is a prospective, randomized, controlled interventional study. Forty participants with mild-to-moderate bruxism or TMJ dysfunction will be randomly assigned to one of two groups:

MODJAW group (n=20): Participants will receive a patient-specific occlusal splint designed based on 3D mandibular kinematic data collected with MODJAW.

Standard splint group (n=20): Participants will receive a conventional occlusal splint fabricated using standard methods.

The study duration for each participant is 8 weeks, during which participants will wear their assigned splints according to instructions and attend follow-up assessments.

Inclusion Criteria:

Age 18-50 years

Diagnosed with mild-to-moderate bruxism or TMJ dysfunction

Willingness and ability to comply with splint use and study visits

Signed informed consent

Exclusion Criteria:

Severe dental loss or existing prosthetic devices interfering with splint placement

Systemic medical conditions affecting jaw function

History of TMJ trauma or surgery

Pregnancy or breastfeeding

Allergy to splint materials

Study Procedures:

Screening and Baseline Assessment:

Clinical examination of dentition and TMJ

Recording baseline jaw movements using MODJAW (for both groups)

Baseline assessment of bruxism frequency, TMJ pain (VAS score), and patient-reported comfort

Splint Fabrication:

MODJAW group: CAD/CAM splints designed using mandibular movement data captured by MODJAW

Standard group: Conventional splints fabricated according to standard occlusal design

Splint Use:

Participants instructed to wear splints nightly (or as directed) for 8 weeks

Weekly check-ins to monitor compliance and comfort

Follow-Up Assessments (Week 4 and Week 8):

Repeat MODJAW recordings to evaluate changes in mandibular movement

Assess TMJ pain, bruxism frequency and intensity

Collect patient satisfaction and comfort scores via 5-point Likert scale

Record any adverse events

Outcome Measures:

Primary Outcome: Changes in mandibular movement patterns as measured by MODJAW

Secondary Outcomes:

Reduction in TMJ pain (VAS score)

Patient-reported satisfaction and comfort

Data Analysis:

Within-group comparisons: Paired t-tests or Wilcoxon signed-rank tests

Between-group comparisons: Mann-Whitney U test

Categorical outcomes: Chi-square or Fisher's exact test

Statistical significance set at p < 0.05

Safety Considerations:

Participants monitored for adverse events related to splint use, including discomfort, tissue irritation, or allergic reactions

Participants may withdraw at any time

All data handled according to confidentiality and privacy guidelines

Significance:

This study will provide evidence on the effectiveness of patient-specific, MODJAW-guided occlusal splints in improving jaw function, reducing bruxism, and increasing patient satisfaction. The results may support the adoption of kinematic data in routine occlusal splint design and contribute to personalized dentistry approaches.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Diagnosed with mild-to-moderate bruxism or temporomandibular joint (TMJ) dysfunction
* Willingness and ability to comply with splint use and study visits
* Signed informed consent

Exclusion Criteria:

* Severe dental loss or existing prosthetic devices interfering with splint placement
* Systemic medical conditions affecting jaw function
* History of TMJ trauma or surgery
* Pregnancy or breastfeeding
* Allergy to splint materials

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-10-15 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-25 (Actual)

PRIMARY OUTCOMES:
Improvement in mandibular movement patterns | Baseline and after 8 weeks of splint use
  Mandibular movements will be recorded using MODJAW 3D jaw-tracking system.
  Parameters include opening, lateral, and protrusive excursions, as well as path stability and range of motion.
  The primary analysis will compare baseline mandibular kinematics to post-intervention measurements between the MODJAW-based splint group and the standard splint group.

SECONDARY OUTCOMES:
TMJ pain levels | Baseline and after 8 weeks of splint use
  Patients pain levels will be assessed using a Visual Analog Scale (VAS).
Comfort and satisfaction | Baseline and after 8 weeks of splint use
  Patient comfort and satisfaction will be assessed using a patient-reported questionnaire and 5-point Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul university, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data (IPD) from this study will not be shared. The study involves patient-specific dental records and intraoral imaging that are considered sensitive and personally identifiable. To protect participant privacy and comply with ethical standards, raw data containing personal identifiers will remain confidential and will not be made publicly available. Aggregate or de-identified summary data may be shared upon reasonable request with qualified researchers following approval from the study team and institutional review board.

REFERENCES:
- See also: Participants will wear their assigned splints for 8 weeks, following study instructions. Outcomes will be assessed at baseline and at the end of the 8-week period. Primary outcomes include improvement in mandibular movement patterns measured using MODJAW — https://pubmed.ncbi.nlm.nih.gov/38945794/